CLINICAL TRIAL: NCT00609739
Title: Cytosine Arabinoside and Mitoxantrone for Patients With Juvenile Myelomonocytic Leukemia Receiving Repeat Stem Cell Transplantation
Status: Terminated | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: Low accrual
Sponsor: Masonic Cancer Center, University of Minnesota (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 1999LS032; UMN-MT1999-08 (Other: Blood and Marrow Transplantation Program); 9906M07303 (Other: IRB, University of Minnesota)
Record Dates: First submitted 2008-02-06; First posted 2008-02-07 (Estimated); Results first posted 2012-03-02 (Estimated); Last update posted 2017-12-28 (Actual); Status verified 2017-12

CONDITIONS: Leukemia
Keywords: juvenile myelomonocytic leukemia
MeSH Terms: conditions — Leukemia; Leukemia, Myelomonocytic, Juvenile | interventions — Cyclosporine; Cytarabine; Filgrastim; Granulocyte Colony-Stimulating Factor; Methotrexate; Methylprednisolone; Mitoxantrone; Cord Blood Stem Cell Transplantation; Isotretinoin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Cytarabine + Mitoxantrone (Experimental): This is a phase I-II study designed to evaluate the efficacy of the administration of high dose cytosine arabinoside and mitoxantrone followed by HCT in patients with JMML who have residual disease or have relapsed after initial HCT.
  Interventions: Drug: cyclosporine; Drug: cytarabine; Drug: filgrastim; Drug: methotrexate; Drug: methylprednisolone; Drug: mitoxantrone hydrochloride; Procedure: allogeneic bone marrow transplantation; Procedure: umbilical cord blood transplantation; Drug: Cis-Retinoic acid

INTERVENTIONS:
Drug: cyclosporine — Patients will receive CSA therapy beginning on day -3, with a taper commencing on day +60 (unless GVHD) and ending on day +90. For patients >40 kg with normal renal function (creatinine <1.3 mg/dL), the initial dose will be 2.5 mg/kg intravenously (IV) over 2 hours every 12 hours. For children <40 kg, the initial dose will be 2.5 mg/kg IV over 2 hours every 8 hours.
  Other Names: CSA
Drug: cytarabine — 3000 mg/m^2 intravenously (IV) over 2 hours x 2 (i.e. total 6000 mg/m^2/day) on days -9 through -4.
  Other Names: Ara-C
Drug: filgrastim — Patients with absolute neutrophil count (ANC) <0.2 x 10^8/L on day 21 may receive G-CSF at 5 mcg/kg/day. G-CSF will be continued until ANC ≥2.5 x 10^8/L for two consecutive days. As the malignant cell population of JMML is known to be hypersensitive to GM-CSF, this cytokine will not be given to these patients.
  Other Names: G-CSF
Drug: methotrexate — MTX will be administered to recipients of non-genotypically identical BMT. MTX will be administered at a dose of 15 mg/m^2 (based on adjusted ideal body weight) intravenously (IV) on day +1 and at a dose of 10 mg/m^2 IV on days +3, +6, and +11.
  Other Names: MTX
Drug: methylprednisolone — Recipients of UCB will receive methylprednisolone 2 mg/kg/day from day +5 to +19 at a dose of 1 mg/kg twice a day (bid) with a 10% taper every week thereafter.
  Other Names: Medrol
Drug: mitoxantrone hydrochloride — 10 mg/m^2 over 30 minutes intravenously (IV) on days -9 through -7.
  Other Names: Mitoxantrone
Procedure: allogeneic bone marrow transplantation — Donor marrow will be collected in the usual sterile manner with a collection goal of 2.0 >10^8/kg recipient weight. Infused on Day 0.
Procedure: umbilical cord blood transplantation — Umbilical cord blood (UCB) will be cryopreserved prior to transplantation. Cord blood units will be selected for transplantation according to current University of Minnesota Department of Blood and Marrow Transplantation Guidelines.
Drug: Cis-Retinoic acid — Post-Transplant Cis-Retinoic Acid (CRA) Therapy - CRA will be given at a dosage of 100 mg/m^2/day by mouth in a single daily dose starting on day +60 and continuing until 1 year after transplant.
  Other Names: isotretinoin

SUMMARY:
RATIONALE: Giving chemotherapy drugs, such as cytarabine and mitoxantrone, before a donor stem cell transplant helps stop the growth of cancer cells and helps stop the patient's immune system from rejecting the donor's stem cells. When certain stem cells from a donor are infused into the patient they may help the patient's bone marrow make stem cells, red blood cells, white blood cells, and platelets. Sometimes the transplanted cells from a donor can make an immune response against the body's normal cells. Giving cyclosporine, methotrexate, and methylprednisolone before or after transplant may stop this from happening.

PURPOSE: This phase I/II trial is studying the side effects and best way to give high-dose cytarabine together with mitoxantrone in treating patients with juvenile myelomonocytic leukemia undergoing a second donor stem cell transplant.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* To determine the incidence of 1-year disease-free survival in patients with juvenile myelomonocytic leukemia and who is undergoing a repeat stem cell transplantation.

Secondary

* To evaluate the incidence of regimen-related toxicity.
* To evaluate the incidence of acute and chronic graft-versus-host-disease.
* To evaluate the incidence of relapse.

OUTLINE:

* Preparative cytoreductive therapy: Patients receive high-dose cytarabine IV over 2 hours on days -9 to -4 and mitoxantrone hydrochloride IV over 30 minutes on days -9 to -7.
* Allogeneic hematopoietic stem cell transplantation (HSCT): Patients undergo HSCT on day 0. Patients undergoing umbilical cord blood transplantation receive methylprednisolone (as graft failure prophylaxis) IV twice daily on days 5 to 19 followed by a taper every other day thereafter until day 25.
* Graft-versus-host-disease (GVHD) prophylaxis: Patients receive cyclosporine IV over 2 hours every 8-12 hours or orally twice daily beginning on day -3 and continuing until day 50, followed by a taper to day 90, in the absence of GVHD. Patients undergoing nongenotypically identical bone marrow transplantation also receive methotrexate IV on day 1 beginning 24 hours after completion of stem cell infusion and on days 3, 6, and 11.
* Post-transplantation isotretinoin therapy: Patients receive oral isotretinoin once daily beginning on day 60 and continuing until 1 year after HSCT.

Patients undergo bone marrow sample collection on day 21, day 60, day 100, at 6 months, and at 1 year for chimerism studies. Patients also undergo blood sample collection periodically to monitor peripheral blood counts for immune reconstitution.

After completion of study treatment, patients are followed on day 21, day 100, at 6 months, and at 1 year.

ELIGIBILITY:
Inclusion Criteria:

* Patients age 0-18 with juvenile myelomonocytic leukemia (JMML) who have relapsed or have residual disease after allogeneic HCT. Residual disease is defined as failure to eradicate original disease without prior documentation of remission. Relapse is defined as reappearance of i) leukocytosis with absolute monocytosis >1 x 10^8/L, ii) presence of immature myeloid cells in the peripheral circulation in two consecutive bone marrow specimens taken at least one month apart, or iii) presence of clonal cytogenetic abnormality. The diagnosis of relapse will be supported by the return of an abnormal cytogenetic marker (if present at diagnosis) or the presence of host cells by RFLP or other method.
* Patients should be at least 6 months from first hematopoietic cell transplant (HCT) if clinically stable. (If JMML is rapidly progressive, second HCT may be performed earlier).

  * Adequate major organ function including:

    * Cardiac: ejection fraction ≥45%
    * Pulmonary: FEV >50%, DLCO >50%
  * Renal: creatinine clearance ≥40 mL/min

    * Hepatic: no clinical evidence of hepatic failure (e.g. coagulopathy, ascites)
  * Karnofsky performance status ≥70% or Lansky score ≥50%
* Written informed consent.

Exclusion Criteria:

* Active uncontrolled infection within one week of HCT.

Max Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 1 (Actual)
Dates: Start 1999-06; Primary Completion 2010-06 (Actual); Study Completion 2010-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Margaret L. MacMillan, MD, Principal Investigator — Masonic Cancer Center, University of Minnesota
Locations (1):
- Masonic Cancer Center at University of Minnesota, Minneapolis, Minnesota, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Only 1 patient was enrolled (yr 1999) and later died (yr 2000). Study was terminated due to low accrual.
Groups:
- Cytarabine + Mitoxantrone: Patients receive administration of high dose cytosine arabinoside and mitoxantrone followed by hematopoietic cell transplant.
Period: Overall Study
Arm/Group | Cytarabine + Mitoxantrone
Started | 1
Completed | 1
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Cytarabine + Mitoxantrone
Number analyzed (Participants) | 1
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 1
  Between 18 and 65 years | 0
  >=65 years | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1
  Male | 0
Region of Enrollment [Number; unit: participants]
  United States | 1

OUTCOME MEASURES:

1. Primary Outcome: Disease-free Survival
Description: Number of patients who were free of disease and alive at 1 year.
Time Frame: 1 year
Measure: Number; unit: Participants
Arm/Group | Cytarabine + Mitoxantrone
Number analyzed (Participants) | 1
Participants | 0

2. Secondary Outcome: Patients With Regimen-Related Toxicity
Description: Number of patients with adverse events related to treatment.
Time Frame: Up to 30 Days Post Study Treatment
Measure: Number; unit: participants
Arm/Group | Cytarabine + Mitoxantrone
Number analyzed (Participants) | 1
participants | 0

3. Secondary Outcome: Patients With Graft-Versus-Host-Disease
Description: Number of patients who exhibited acute and/or chronic graft-versus-host disease.
Time Frame: Up to 30 Days Post Study Treatment
Measure: Number; unit: participants
Arm/Group | Cytarabine + Mitoxantrone
Number analyzed (Participants) | 1
participants | 1

4. Secondary Outcome: Patients Who Relapsed
Description: Number of patients whose disease relapsed.
Time Frame: 1 Year
Measure: Number; unit: participants
Arm/Group | Cytarabine + Mitoxantrone
Number analyzed (Participants) | 1
participants | 1

ADVERSE EVENTS:
Time Frame: Up to 30 days post study treatment.
Description: Regimen related toxicity (RRT) is a concern, but because of the seriousness of relapsed JMML, a high incidence of grade III and IV RRT will be considered acceptable. No other adverse events were collected.
Arm/Group | Cytarabine + Mitoxantrone
Serious Adverse Events (participants affected / at risk) | 1/1
Other Adverse Events (participants affected / at risk) | 0/1
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Cytarabine + Mitoxantrone (N=1)
Death (General disorders) | 1 (1)

LIMITATIONS AND CAVEATS:
Only 1 patient was enrolled (yr 1999) and later died (yr 2000). Study was terminated due to low accrual.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes